CLINICAL TRIAL: NCT00178971
Title: Serotonin 1A Agonists and Cognition in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Herbert Meltzer, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 020724
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): buspirone 15-30 mg qd
  Interventions: Drug: adjunctive treatment with buspirone
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: adjunctive treatment with buspirone — buspirone 15-30 mg qd
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
Examines cognitive functioning in patients with schizophrenia or schizoaffective disorder who have been treated with antipsychotic medications. Patients will be assigned to take active medication (Buspar)or placebo along with their prescribed antipsychotic medication for six weeks. Patients' memory and problem-solving ability will be tested before and after medication.

DETAILED DESCRIPTION:
Examines cognitive functioning in patients with schizophrenia or schizoaffective disorder who have been treated with olanzapine or risperidone for at least three months randomized to receive adjunctive treatment with a 5-HT1A agonist (buspirone, 15-30 mg/day)or placebo.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for participation in the current research study.

1. Subjects will be males and females between 18-65 years of age;
2. Subjects will have a definite diagnosis by DSM-IV criteria for Schizophrenia or Schizoaffective Disorder;
3. The subjects or their legal guardian must sign the informed consent;
4. Subjects currently being treated with olanzapine or risperidone for a duration of at least 3 months

Exclusion Criteria:

1. Subjects who are pregnant or lactating
2. Subjects who have brain damage and/or neurological disorders
3. Subjects who have current substance dependence
4. Subjects unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-01; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
This study will examine the effect on cognition of the addition of buspirone compared with addition of a sugar pill to patients treated with olanzapine or risperidone | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Y Meltzer, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Psychiatric Hospital at Vanderbilt, Nashville, Tennessee, United States